CLINICAL TRIAL: NCT00078533
Title: Virus Specific Cytotoxic T-Lymphocytes for the Treatment of CMV After Allogeneic Stem Cell Transplant: A Dose-Finding Trial
Brief Title: Cytotoxic T-Lymphocytes for the Prophylaxis of Cytomegalovirus After Allogeneic Stem Cell Transplant
Acronym: VICTA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Helen Heslop, Professor of Medicine and Pediatrics, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12683-VICTA; VICTA (Other: Baylor College of Medicine); PACT 001 (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2004-03-01; First posted 2004-03-02 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-06

CONDITIONS: Cytomegalovirus Infections
Keywords: Allogeneic; Transplant; CMV; Stem Cell; Donor; Allogeneic stem cell recipients at risk for CMV reactivation
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CMV CTL infusion (Experimental): Subjects are assigned a dose level at the time of enrollment.
  Interventions: Biological: CMV CTL infusion

INTERVENTIONS:
Biological: CMV CTL infusion — Three dose levels will be explored. The lowest dose level will be 1x10^7cells/m2 and the highest will be 1x10^8/m2. 3-6 pts will be entered at each dose level (depending on toxicity). If there are no toxicities and immunological efficacy is not seen at any dose, then the doses will be further escalated after additional local and federal approval. Additional patients will be treated at dose level 1 in order to assess the secondary objective of virus-specific immunity from the CTL infusions

SUMMARY:
Patients have a type of blood cell cancer, other blood disease or a genetic disease for which they will receive a stem cell transplant. The donor of the stem cells will be either a brother or sister or another relative or a closely matched unrelated donor. We are asking patients to participate in this study which tests if blood cells from the donor that have been grown in a special way, can prevent the patients from getting an infection with a virus called Cytomegalovirus or CMV.

CMV is a virus that can cause serious infections in patients with suppressed immune systems. It usually affects the lungs and can cause a very serious pneumonia, but it can also affect the intestinal tract, the liver and the eyes. Approximately 2/3 of normal people harbor this virus in their body. In healthy people CMV rarely causes any problems because the immune system can keep it under control. If the patient and/or their donor is positive for CMV, they are at risk of developing CMV disease while the patients immune system is weak post transplant. Usually, this risk is highest during the first 3-4 months after the transplant.

CMV disease can be prevented during this time in most people by using drugs that can kill the virus such as Ganciclovir, Foscarnet, or Cidofovir . However, these medications have many side effects and have to be given daily by vein for approximately 4-5 months after transplant. One of the side effects is that it takes the new immune system much longer to develop an effective defense against the virus. Therefore, once the medicines are stopped, the patients still have a chance to develop CMV disease.

We want to see if we can use a kind of white blood cell called T cells that we have grown from the stem cell donor instead of the regular treatment with Ganciclovir or Foscarnet to prevent CMV from "flaring up". These cells have been trained to attack CMV virus infected cells. We will grow these T cells from blood taken from the donor before the patients transplant. These cells are called CMV-specific cytotoxic T-lymphocytes or CMV CTL, and they will be given to the patient around 30 days after their transplant.

We have used this sort of therapy to treat a different virus which can cause problems after transplant called Epstein Barr Virus (EBV). Doctors at other places have used similar T cells to treat or prevent CMV infections after transplant and have not seen any significant problems. These CMV specific cytotoxic T cells are an investigational product not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
If the patient and their donor are eligible, we will take 100-120 ml (20-24 teaspoonfuls) of blood from the donor 3-4 weeks before the transplant. We will only take as much blood as is safe for the patient and their donor.

We will use this blood to grow T cells. We will first infect the peripheral blood mononuclear cells with a specially produced human virus adenovirus) that carries part of the CMV gene to the monocytes which will stimulate the T cells. This stimulation will train the T cells to kill cells with the pp65 from the CMV virus on their surface. If this approach is insufficient to stimulate T cells which will kill the pp65 from the CMV virus then we will grow a special type of cell called dendritic cells which will stimulate the T cells and we will put the specially produced human virus (adenovirus) that carries the parts of the CMV gene (called pp65) into the dendritic cells. These dendritic cells will then be treated with radiation so they cannot grow. They will then be used to stimulate T cells. This stimulation will train the T cells to kill cells with the pp65 from the CMV virus on their surface.

We will then grow these CMV specific CTLs by more stimulation with EBV infected cells (which we will make from the blood of the donor by infecting them with EBV in the laboratory). We will also put the adenovirus that carries the CMV pp65 gene into these EBV infected cells so that they too have CMVpp65. These EBV infected cells will be treated with radiation so they cannot grow. Once we have made sufficient numbers of T cells we will test them to make sure they kill cells with CMVpp65 on their surface. To make sure that these cells won't attack the patients tissues, we test these cells against the lymphoblasts that we grow in the laboratory. These will be used to check if the CMV CTL can attack them. Alternatively, we could take a small piece of skin from the patient to grow skin cells which can also be used to check if CMV CTL can attack them. The skin biopsy can be done at the same time of another procedure such as a bone marrow.

The donor's CMV CTL cells will be thawed and injected into the patients intravenous line for a period of 10 minutes after the patient received Benadryl and Tylenol. The patient will receive the dose of CMV CTL cells on or after day 30 following their transplant if they agree and are well enough. We will not give antiviral medications during this study but we will monitor the CMV levels weekly for at least 30 days after the transplant. If after the initial dose of CMV CTL cells the patient develops a viral infection, then they may be eligible to receive one additional injection of CTLs at the same dose as the first injection. If the CMV levels in the blood continue to rise after the dose of T cells then the patient will receive treatment with Ganciclovir, Foscarnet, or Cidofuvir.

The patient will continue to be followed in the BMT clinic after the injection. They will be seen in the clinic, in the hospital or contacted by the research nurse and have blood tests (to monitor the blood counts, the kidney and liver function and to monitor for viruses) weekly for the first 60 days after the CTL infusion, then at 3, 6, 9 and 12 months. To learn more about the way the T cells are working in the body, an extra 20-40 mls (4-8 teaspoons) of blood will be taken before the infusion and then 24 hours after the infusion (optional depending on the patients preference), and then at 1, 2, 4 and 6 weeks after the infusion. After this, blood will be taken every 3 months for 1 year. The amount of blood taken in the first 12 months will be 260-460mls (1-2 cups). Total time participation for this study will be 1 year.

ELIGIBILITY:
Inclusion criteria:

* Recipients of allogeneic donor stem cell transplants at risk for CMV reactivation with a CMV seropositive stem cell donor and at least 30 days post transplant.
* Recipients can have early evidence of CMV reactivation with greater than 2 leukocytes but less than 10 leukocytes positive for the CMV Ag per 100,000 cells.
* No evidence of graft-versus-host disease (GVHD) > Grade II at time of enrollment.
* Life expectancy > 30 days
* No severe intercurrent infections
* Lansky/Karnofsky scores greater than or equal to 60
* Absence of severe renal disease (Creatinine > x 3 normal for age)
* Absence of severe hepatic disease (direct bilirubin > 3 mg/dl or SGOT > 500)
* Not receiving Ganciclovir, Foscarnet, or Cidofovir or other antiviral therapy for CMV reactivation
* Patient/guardian able to give informed consent

Exclusion Criteria:

* Patients with CMV negative stem cell donors
* Patients with GVHD Grades III-IV
* Patients receiving antiviral therapy for CMV reactivation or other viral infections such as adenovirus or herpes viruses
* Patients with significant CMV reactivation. Significant CMV reactivation is defined as one CMV Antigenemia reading with >10 leukocytes positive for the CMV Ag per 100,000 cells
* Patients with less than 50% donor chimerism in either peripheral blood or bone marrow or patients with relapse of original disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-04; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
safety, toxicity and maximum tolerated dose (MTD) | 30 days
Efficacy of recovery of virus-specific immunity and correlation with protection from viral reactivation/disease. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Keller MD, Darko S, Lang H, Ransier A, Lazarski CA, Wang Y, Hanley PJ, Davila BJ, Heimall JR, Ambinder RF, Barrett AJ, Rooney CM, Heslop HE, Douek DC, Bollard CM. T-cell receptor sequencing demonstrates persistence of virus-specific T cells after antiviral immunotherapy. Br J Haematol. 2019 Oct;187(2):206-218. doi: 10.1111/bjh.16053. Epub 2019 Jun 20. PMID 31219185
- [Derived] Hanley PJ, Cruz CR, Savoldo B, Leen AM, Stanojevic M, Khalil M, Decker W, Molldrem JJ, Liu H, Gee AP, Rooney CM, Heslop HE, Dotti G, Brenner MK, Shpall EJ, Bollard CM. Functionally active virus-specific T cells that target CMV, adenovirus, and EBV can be expanded from naive T-cell populations in cord blood and will target a range of viral epitopes. Blood. 2009 Aug 27;114(9):1958-67. doi: 10.1182/blood-2009-03-213256. Epub 2009 May 14. PMID 19443656